CLINICAL TRIAL: NCT05898074
Title: Novel Application of RADA16 Hydrogel in Reducing Sinonasal Morbidity After Endoscopic Skull Base Surgery
Brief Title: Role of Novel RADA16 Hydrogel in Endoscopic Skull Base Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: 3-D Matrix UK Ltd. (Industry)
Responsible Party: Principal Investigator, Satyan B. Sreenath, Assistant Professor, Department of Otolaryngology--Head and Neck Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14045
Record Dates: First submitted 2023-05-22; First posted 2023-06-12 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Skull Base Neoplasms; Cerebrospinal Fluid Leakage; Nasal; Hypertrophy, Mucous Membrane (Septum)
Keywords: Nasoseptal Flap Harvest; Sinonasal Morbidity; Extracellular Matrix; Endoscopic Skull Base Surgery
MeSH Terms: conditions — Skull Base Neoplasms; Cerebrospinal Fluid Leak; Hypertrophy

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized Cohort Study
Who Masked: Outcomes Assessor
Masking Description: This will be double blinded (video endoscopy will be performed and scoring will be performed by non-operative surgeon, blinded to the intervention group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PuraGel (RADA16) Hydrogel (Active Comparator): Participant will have PuraGel (RADA16) Hydrogel applied to the nasoseptal flap harvest site following endoscopic skull base surgery
  Interventions: Device: PuraGel (RADA16) Hydrogel
- Non-absorbable Packing (Silastic Splint) (Active Comparator): Participant will have a silastic splint (Non-Absorbable Packing) applied to the nasoseptal flap harvest site following endoscopic skull base surgery with no additional packing or agent
  Interventions: Device: Non-Absorbable Packing (Silastic Splint)

INTERVENTIONS:
Device: Non-Absorbable Packing (Silastic Splint) — Participant will have silastic splint applied to nasoseptal flap harvest site
  Arms: Non-absorbable Packing (Silastic Splint)
Device: PuraGel (RADA16) Hydrogel — Participant will have PuraGel (RADA16) Hydrogel applied to the nasoseptal flap harvest site
  Arms: PuraGel (RADA16) Hydrogel

SUMMARY:
The purpose of this study is to specifically evaluate the effectiveness of PuraGel, a RADA16 polypeptide hydrogel, in expediting post-operative healing and re-mucosalization of the nasoseptal flap harvest site during endoscopic skull base surgery and the impact on patient and sinonasal morbidity.

DETAILED DESCRIPTION:
Briefly, multiple agents exist and have been long-studied in endoscopic sinus and septal surgery, which include non-absorbable agents and biodegradable, absorbable synthetic agents including extracellular matrix (ECM) based compounds and synthetic biopolymers. The goal of these agents has often been to reduce sinonasal crusting, postoperative bleeding, and synechia formation. With advancements in postoperative adjuncts, many options now exist for postoperative sinonasal packing including medicated products such as steroid-impregnated stents and chitosan-based absorbable packs.

Lastly, with respect to intra-operative adjuncts designed to foster healing in the postoperative period, PuraGel, a RADA16 polypeptide hydrogel, was identified as an ECM-based solution, which aids in wound healing, adhesion prevention, and hemostasis at the completion of the case. In hydrogel format, this agent forms a synthetic matrix that serves as a scaffold for mucosal healing while serving as a mechanical barrier on tissue surfaces, thereby limiting scarring. To date, there have been no studies evaluating the role of this gel-based compound in the postoperative period in endoscopic skull base surgery.

Thus, amongst all of these agents that have been previously studied to some degree in patients undergoing endoscopic sinus surgery, there has been limited study on their role in endoscopic skull base surgery and utility in reducing sinonasal morbidity in the postoperative setting. Therefore, our goal was to investigate and compare the impact of varying sinonasal agents in the nasal cavity following endoscopic skull base surgery. We hypothesize that the absorbable, ECM-based gel compound (PuraGel) demonstrates an improvement on postoperative healing rate and sinonasal crusting with reduced patient morbidity and improved patient comfort when compared to non-absorbable agents.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient is undergoing endoscopic endonasal approach for the management of a skull base tumor or cerebrospinal fluid leak. Nasoseptal Flap must be harvested.
* Patient is undergoing surgery via bi-nostril approach requiring bilateral surgical dissection of the nasal cavity in approach to the skull base

Exclusion Criteria:

* Patient has evidence of radiographic baseline sinus disease consistent with acute or chronic rhinosinusitis (including nasal polyposis, prior septal perforation) on pre-operative CT sinus
* Patient has had prior sinonasal surgery or has undergone sinonasal radiation treatment
* Patient has a known coagulation disorder or immune deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-10-09 (Estimated); Study Completion 2025-10-09 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Lund-Kennedy nasal endoscopy score | 1 week, 4 weeks, and 12 weeks following surgery.
  Modified Lund-Kennedy nasal endoscopy score to rate mucosal edema, nasal crusting, and scarring. This will be double blinded (video endoscopy will be performed and scoring will be performed by non-operative surgeon, blinded to the intervention group). This scoring will address wound healing, adhesion formations. Scoring will be performed at 1 week, 4 weeks, and 12 weeks following surgery. The timing of these assessments is based on the routine postoperative follow-up schedule. No additional appointments will be made for the purposes of this study. We will be looking at the change in this score over time.
  Minimum would be 0. Maximum would be 10. Higher score means worse outcome. The un-abbreviated title is Modified Lund-Kennedy nasal endoscopy score.

SECONDARY OUTCOMES:
Patient-reported pain | 1 week, 4 weeks, and 12 weeks following surgery.
  Patient-reported pain visual analog scale during postoperative debridement of the main nasal cavity. Minimum score is 1 (reflecting no pain) and the maximum score is 10 (reflecting extreme amount of pain).
  Minimum would be 0. Maximum would be 10. Higher score means worse outcome. The un-abbreviated title is Patient-reported pain visual analog scale.
subjective QOL score | 1 week, 4 weeks, and 12 weeks following surgery.
  Postoperative, subjective QOL score with the validated Anterior Skull Base Nasal Inventory-12 (ASK-12) at 1 week, 4 weeks, and 12 weeks postoperatively.
  Minimum would be 0. Maximum would be 72. Higher score means worse outcome. The un-abbreviated title is Anterior Skull Base Nasal Inventory-12.
Endoscopic grading of mucosalization | 1 week, 4 weeks, and 12 weeks following surgery.
  Likert scale of mucosalization of the nasal septum graded by blinded reviewer via nasal endoscopy video
  Minimum would be 0. Maximum would be 10. Higher score means worse outcome. The un-abbreviated title is Likert scale of mucosalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No